CLINICAL TRIAL: NCT06776367
Title: Longitudinal Assessment of Potential Immunologic Correlates of Risk and Protection Following COVID-19 Vaccination Comparing Remote and Site-based Specimen Collection (Feasibility, Validity, and Proof of Concept)
Brief Title: Project REMOTE (REimagining Measurements and Operations of Translational Endpoints)
Acronym: REMOTE
Status: Active, not recruiting | Type: Observational
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Collaborators: Fred Hutchinson Cancer Center (Other); Allucent (Unknown)
Responsible Party: Sponsor
Other Study IDs: BP-24-001; 75A50123D00005. (Other Grant/Funding Number: Barda)
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: COVID-19; Pandemic Preparedness; COVID-19 vaccine; immune correlates; self-collected; feasibility
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Peripheral Blood Mononuclear Cells (PBMC), saliva, nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: In-clinic study visits and clinic-collected specimens
  Interventions: Other: Traditional clinical trial participation with clinician-collected specimens
- Group B: Fully remote evaluation and self-collected specimens
  Interventions: Other: Remote study participation and self-collection of specimens

INTERVENTIONS:
Other: Remote study participation and self-collection of specimens — Participants in Group B will complete all study procedures remotely and will not physically visit any clinical research site. This will include telehealth (videoconference) visits with study personnel, self-collection of specimens, shipping of specimens using pre-labeled packaging, and completion of electronic diaries for data collection.
  Groups: Group B
Other: Traditional clinical trial participation with clinician-collected specimens — Participants in Group A will attend study visits in person at a clinical research site and will have the majority of specimens collected by a clinician at the clinic. Group A participants will have some electronic diary usage.
  Groups: Group A

SUMMARY:
This trial is designed to assess immunological biomarkers measured from blood samples that can be used to reliably predict how well vaccines work against symptomatic COVID-19 as well as to evaluate the feasibility of remote, self-collected specimens when conducting a correlates analysis. For a lot of research studies, people need to go to the study doctor's office regularly. For this study, we want to see if it is okay that people do the study doctor visits virtually, fill out questionnaires electronically, and collect their own samples remotely.

Participants will enroll in the study after receiving a COVID-19 vaccine in their community, and saliva and blood specimens will be collected at pre-defined time-points over a 12-month period. Additionally, participants will report weekly whether they experience symptoms of COVID-19, and if so, will be prompted to collect a nasal swab for testing. Most participants will complete all activities remotely and via electronic communications, but a small number will complete activities in person at the doctor's office to provide a comparison group.

Samples from the study will be analyzed to determine whether the biomarkers can be measured, and data from the study will be used to evaluate the feasibility of doing the specimen and data collection without the participant going to the doctor's office in person.

DETAILED DESCRIPTION:
This is a non-interventional, minimal-risk, observational study to determine correlates of an FDA-authorized/approved COVID-19 vaccine in a heterogeneous US population. Most participants will be remotely consented, screened, enrolled, and randomized outside of a physical clinical research site. Participants will be screened for study participation from Days -14 to -1 either remotely or at a clinical research site. After screening, eligible participants will be enrolled and will be randomized to one of two groups. Participants randomized to Group A (n~200) will be evaluated at a traditional clinical research site to include site visits for venous blood and saliva specimens to be collected by appropriately trained site personnel within 7 days of enrollment and again at approximately Months 1, 3, 6 and 12. Participants randomized to Group B (n~3800) will undergo fully remote evaluation to include self-collection of capillary blood and saliva specimens occurring within 7 days of enrollment, after receipt of the self-collection sample kits/wearable device. Self-collection will be aided by the electronic Clinical Outcome Assessment (eCOA) platform and/or virtual telehealth visits with the site staff and will occur within 7 days of enrollment and approximately at Months 1, 3, 6, and 12 to mirror group A visits.

Though not part of the study, participants will be required to obtain a currently FDA-approved or -authorized COVID-19 vaccine as part of the inclusion criteria. Participants will be followed for 12 months from receipt of vaccination. Both groups will be surveilled with weekly queries for COVID-19 like symptoms for the duration of the study using an eCOA application on the participant's tablet or smartphone. Should Group A participants identify the presence of COVID-19 like symptoms they will be prompted to schedule an acute visit with their respective site where site staff will collect a nasal swab for PCR to confirm COVID-19 disease. Should Group B participants identify the presence of COVID-19 like symptoms they will be prompted to schedule an acute telehealth visit with their respective site and then self-collect a nasal swab for PCR to confirm COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Are willing and able to provide voluntary electronic informed consent (eConsent) to participate in the study and written authorization (via electronic signature) for use and disclosure of protected health information
* Are able to understand and comply with planned study procedures, including specimen collection devices, use of eCOA application on a tablet or smartphone, and the wearable biometric device.
* Are ≥18 years old at time of informed consent
* Are available for all study data collection timepoints
* Completed primary approved/authorized COVID-19 vaccination series, defined as previous receipt of one of the following options:

  * Doses of original monovalent mRNA or bivalent mRNA vaccine or a combination of the two,
  * Doses of original monovalent Novavax COVID-19 Vaccine, alone or in combination with any mRNA vaccine doses; or
  * Doses of Janssen COVID-19 Vaccine, alone or in combination with any mRNA or Original monovalent Novavax vaccine doses.
* Receipt of an FDA licensed/authorized COVID-19 vaccine within the previous 14 days or on the day of enrollment

Exclusion Criteria:

* Receipt or planned receipt of any of the following vaccines, on the same day or within 28 days prior to or after receipt of the FDA licensed/authorized COVID-19 vaccine:

  * Shingrix (Zoster Vaccine Recombinant, Adjuvanted)
* Receipt of COVID-19 vaccine within 120 days prior to current vaccine
* Any disease or medical condition that, in the opinion of the Investigator or appropriate sub-investigator, is a contraindication to study participation
* Pregnant individuals (only exclusionary for the peripheral blood mononuclear cells [PBMCs] blood draws portion of the study)
* Currently participating or plans to participate in another clinical trial that is interventional and/or involving an investigational product.
* Are assessed by the Investigator as unsuitable for participation in this study for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population: approximately 4,000 individuals in the US with the following considerations:
  * Target 25% of participants ≥65 years of age
  * Appropriate representation of participants at high risk for severe COVID-19
  * Appropriate representation of racially and ethnically diverse populations
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Determine correlates of risk and protection of an FDA-authorized/approved COVID-19 vaccine in a heterogeneous US population using self-collected specimens (Group B only) | From Enrollment through Day 366
  Serum S protein-specific binding antibody (bAb) concentrations (peak and exposure-proximal assessments)
  * Serum SARS-CoV-2 specific neutralizing antibody (nAb) titers (peak and exposure-proximal assessments)
  * COVID-19: Virologically confirmed SARS-CoV-2 infection (by qualitative reverse transcriptase polymer chain reaction [PCR]), along with one or more of the following: fever, chills, cough, headache, fatigue, diarrhea, new loss of taste or smell, sore throat, congestion, runny nose, nausea or vomiting, shortness of breath or difficulty breathing, or muscle or body ache

SECONDARY OUTCOMES:
Determine correlates of risk and protection of an FDA-authorized/approved COVID-19 vaccine in a heterogeneous US population (across Groups A and B) | From Enrollment through Day 366
  Serum S protein-specific binding antibody (bAb) concentrations (peak and exposure-proximal assessments)
  * Serum SARS-CoV-2 specific neutralizing (nAb) antibody titers (peak and exposure-proximal assessments)
  * COVID-19: Virologically confirmed SARS-CoV-2 infection (by qualitative reverse transcriptase polymer chain reaction [PCR]), along with one or more of the following: fever, chills, cough, headache, fatigue, diarrhea, new loss of taste or smell, sore throat, congestion, runny nose, nausea or vomiting, shortness of breath or difficulty breathing, or muscle or body ache.
Determine correlates of risk and protection of an FDA-authorized/approved COVID-19 vaccine against severe disease in a heterogeneous US population (Group B only) | From Enrollment through Day 366
  Serum S protein-specific bAb concentrations (peak and exposure-proximal assessments)
  * Serum SARS-CoV-2 specific nAb titers (peak and exposure-proximal assessments)
  * COVID-19 per Primary Objective Endpoint definition, plus any one or more of the following: clinical signs indicative of severe systemic illness, respiratory Rate ≥ 30 per minute, heart rate ≥ 125 beats per minute, SpO2 ≤ 93% on room air at sea level or PaO2/FIO2 < 300 mm Hg, respiratory failure or Acute Respiratory Distress Syndrome (ARDS)1, evidence of shock2, significant acute renal, hepatic, or neurologic dysfunction, admission to an intensive care unit or death
Assess the feasibility of gathering valid remote self-collected specimens (across Groups A and B) | From Enrollment through Day 366
  Number of self-collected nasal swabs, saliva specimens, and capillary blood specimens received vs expected
  * Comparison of proportion of valid specimens among self-collected capillary blood specimens to clinical-site venous specimens
  * Acceptability and tolerance of specimen collection methods
Assess safety of an FDA authorized/approved COVID-19 vaccine (across Groups A and B) | From Enrollment through Day 181
  Serious adverse events (SAEs) through 6 months following vaccination

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Accel Research Site Networks - Birmingham CRU / Elite, Vestavia Hills, Alabama
  - Desert Clinical Research, Mesa, Arizona
  - Apex Research Group, Fair Oaks, California
  - Wake Research Encino, Los Angeles, California
  - Wake Research San Diego, San Diego, California
  - Research Institute of South Florida, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Wake Research Atlanta, Atlanta, Georgia
  - Johnson County Clinical Trials (JCCT), Lenexa, Kansas
  - Research Integrity / WCG, Owensboro, Kentucky
  - Alcanza / hyperCORE, Boston, Massachusetts
  - Be Well Clinical Studies / Elite, Lincoln, Nebraska
  - SUNY / Upstate Medical University Global Health Institute, Syracuse, New York
  - Kroger The Little Clinic (Remote Site), Blue Ash, Ohio
  - Lynn Health Science Institute East / Elite, Oklahoma City, Oklahoma
  - Wake Research Dallas, Dallas, Texas